CLINICAL TRIAL: NCT07046195
Title: Clinical Study of the Optimal Combination Mode of Adjuvant Radiotherapy Combined With Immunotherapy for Triple Negative Breast Cancer
Brief Title: Optimal Combination of Adjuvant Radiotherapy and Immunotherapy for Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023ZD0502302
Record Dates: First submitted 2025-06-09; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Hypofractionated Radiotherapy; Triple Negative Breast Cancer (TNBC); Immunotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Concurrent group: Patients receiving concurrent immunotherapy, that is, at least 1 dose of immunotherapy between 1 week before radiotherapy and the end of radiotherapy
- Sequential group: Patients receiving sequential immunotherapy, that is, 1 week before the start of radiotherapy or 2 weeks after the end of radiotherapy

SUMMARY:
Postoperative radiotherapy is a conventional treatment for breast cancer patients with a high risk of recurrence, such as those with regional lymph node metastasis, especially TNBC. However, the optimal mode of treatment for the combination of radiotherapy and immunotherapy has not yet been determined, especially in the adjuvant treatment phase. There is still a lack of validation and high-grade evidence on the safety and synergistic efficacy of radiotherapy-immunotherapy combinations. In this study, we aimed to compare the safety and preliminary efficacy of hypofractionated radiotherapy and concurrent immunotherapy with those of hypofractionated radiotherapy and sequential immunotherapy in the postoperative adjuvant stage through prospective real-world studies for TNBC patients, and focused on verifying the incidence of adverse reactions in radiotherapy and immunotherapy in the adjuvant stage, so as to find out the optimal combination mode of postoperative radiotherapy combined with immunotherapy, further reduce the distant metastasis of TNBC patients under the premise of ensuring safety, and improve long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. Triple negative invasive breast cancer, with immunohistochemistry confirming that the primary lesion was ER- or ER<10% and weakly expressed, PR-, HER 2-;
3. Patients who had surgery after neoadjuvant immunotherapy, and required a hypofractionated radiotherapy regimen of whole breast/chest wall ± regional lymph nodes ±tumor bed: whole breast/chest wall ± regional lymph nodes DT 40.05Gy/15F; Sequential dose increase of DT 2.9 Gy*3F for tumor bed in breast conserving patients; For patients with a stage of T4 or N3c, it is up to the radiation oncologist to decide whether to proceed with sequential bolsing of locoregional lesions;
4. Patients received adjuvant immunotherapy after neoadjuvant immunotherapy, and the drugs used for postoperative immune maintenance were the immunodrugs used in the neoadjuvant treatment stage;
5. Patients who have not received neoadjuvant immunotherapy and require 1 year of adjuvant immunotherapy and hypofractionated intensity-modulated radiotherapy for whole breast/chest wall ± regional lymph nodes ± tumor beds in the postoperative adjuvant stage.

Exclusion Criteria:

1. Failure to complete the course of radiotherapy as planned
2. Concomitant contralateral breast cancer or second primary malignancy (except basal cell carcinoma of the skin and carcinoma in situ of the cervix);
3. Previous history of thoracic radiotherapy;
4. Serious heart, lung, liver, kidney, hematopoietic and nervous system diseases, mental diseases;
5. Concomitant autoimmune diseases such as scleroderma or active lupus erythematosus; pregnant and lactating patients;
6. Patients with prior immunotherapy-related grade 3-4 toxicities during the neoadjuvant immunotherapy phase

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Tripple negative breast cancer patients who require hypofractionated radiotherapy and immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 adverse reactions | From enrollment to 4 months after the end of treatment
  Treatment-related adverse reactions are defined as those within 120 days of radiotherapy or during and after immunotherapy.

SECONDARY OUTCOMES:
ipsilateral breast tumor recurrence | From date of enrollment, through study completion, an average of 5 years
  Any ipsilateral chest wall, breast recurrence events during the follow-up period
Local-regional Recurrence | From date of enrollment, through study completion, an average of 5 years
  Any ipsilateral chest wall, breast, regional lymph node recurrence event during the follow-up period
Distant metastasis | From date of enrollment, through study completion, an average of 5 years
  Any distant metastasis during the follow-up period.
Distant metastasis free survival | From date of enrollment, through study completion, an average of 5 years
  The time from the date of randomization of the subject to the earliest occurrence of distant metastases or death
Disease free survival | From date of enrollment, through study completion, an average of 5 years
  The time from the date of randomization of the subject to the time of disease recurrence or death of the patient due to disease progression
Overall Survival | From date of enrollment, through study completion, an average of 5 years
  From the date of randomization of the subject to the death of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No